CLINICAL TRIAL: NCT01702545
Title: Determination of Drugs and Their Metabolites in Hospitalized Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Klinikum Nürnberg (Other)
Responsible Party: Principal Investigator, Mr. Prof. Dr. Wilhelm, Prof. Dr. med. Martin Wilhelm, Klinikum Nürnberg
Other Study IDs: PEAK-001
Record Dates: First submitted 2012-10-01; First posted 2012-10-08 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Blood, Plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
The current state of knowledge on the concentration of drugs and their metabolites in the individual human body is not satisfying concerning the question about behavior of drugs in the human body, taking into account individual patient factors such as age, weight and organ dysfunctions.

This projects deals with the question of drug levels in the blood of hospitalized patients.

The aim of this study is to extend the knowledge about the behavior of drugs in the human body significantly, for the safety and benefit of future patients. This also includes to establish a relationship between drug levels in patients and the desired and undesired effects of a drug.

As a result, the future perspective is to find the optimal dose for the individual patient by measuring the blood concentration of a drug.

DETAILED DESCRIPTION:
The primary goal of the study is to gain an overview of the plasma concentrations of relevant drugs which occur in different patient populations and to what extent they are consistent with those concentrations described in the literature.

If the expectation is confirmed, that a significant heterogeneity in the plasma concentrations of these patients exists, the investigators will try to find influencing factors for this circumstance on the basis of routine clinical parameters (height, weight, renal function, concomitant medications, etc.).

Ultimately, this project will identify substances with a high interindividual variability in plasma levels, where drug monitoring might be suggested.

ELIGIBILITY:
Inclusion Criteria:

* legal capacity

Exclusion Criteria:

* severe anemia

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2012-08; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Plasma concentrations [ng/mL] of various drugs at different timepoints | up to five years

CONTACTS AND LOCATIONS:
Overall Officials: Martin Wilhelm, Prof Dr., Study Chair — Paracelsus Medical University Klinikum Nuremberg, Germany
Locations (1):
- Dept. of Internal Medicine V, Klinikum Nürnberg Nord, Nuremberg, Bavaria, Germany